CLINICAL TRIAL: NCT03556293
Title: IMPROVE AKI: A Cluster-Randomized Trial of Team-Based Coaching Interventions to IMPROVE Acute Kidney Injury
Brief Title: IMPROVE AKI Cluster-Randomized Trial
Acronym: IMPROVE-AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Vanderbilt University (Other); University of Vermont (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeremiah R. Brown, Study Contact PI, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: D18114; R01DK113201 (NIH)
Record Dates: First submitted 2018-04-30; First posted 2018-06-14 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Health Planning Technical Assistance

STUDY DESIGN:
Intervention Model Description: 2x2 factorial cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Technical Assistance (No ASR) (Active Comparator): Technical Assistance (TA). Intervention: TA will be offered to the 4 teams randomized to the TA condition without automated surveillance reporting and will receive the AKI Prevention Toolkit plus monthly technical calls independently
  Interventions: Behavioral: AKI Prevention Toolkit; Behavioral: Technical Assistance (TA)
- Virtual Learning Collaborative (No ASR) (Active Comparator): Virtual Learning Collaborative (VLC). Intervention: The VLC will be offered to 4 teams without automated surveillance reportingand will receive the AKI Prevention Toolkit plus monthly virtual training calls with the other VLC sites. Each participating site will be supported to establish a multidisciplinary team charged with continuously improving AKI, which will include interventional cardiologists, cardiac catheterization lab manager and technicians, nursing representatives from the intensive care unit and/or holding areas, cardiology administration, nephrology, and representation from the quality improvement department (VA Clinical Application Coordinator [CAC] and Systems Redesign).
  Interventions: Behavioral: AKI Prevention Toolkit; Behavioral: Virtual Learning Collaborative (VLC)
- Technical Assistance with ASR (Active Comparator): Technical Assistance (TA). Intervention: TA will be offered to the 4 teams randomized to the TA condition with automated surveillance reporting (ASR) and will receive the AKI Prevention Toolkit plus monthly technical calls independently and monthly ASR dashboard.
  Interventions: Behavioral: AKI Prevention Toolkit; Behavioral: Technical Assistance (TA); Behavioral: Automated Surveillance Reporting (ASR)
- Virtual Learning Collaborative with ASR (Active Comparator): Virtual Learning Collaborative (VLC). Intervention: The VLC will be offered to 4 teams with automated surveillance reporting (ASR) and will receive the AKI Prevention Toolkit plus monthly virtual training calls with the other VLC sites with the and monthly ASR dashboard. Each participating site will be supported to establish a multidisciplinary team charged with continuously improving AKI, which will include interventional cardiologists, cardiac catheterization lab manager and technicians, nursing representatives from the intensive care unit and/or holding areas, cardiology administration, nephrology, and representation from the quality improvement department (VA Clinical Application Coordinator [CAC] and Systems Redesign).
  Interventions: Behavioral: AKI Prevention Toolkit; Behavioral: Virtual Learning Collaborative (VLC); Behavioral: Automated Surveillance Reporting (ASR)

INTERVENTIONS:
Behavioral: AKI Prevention Toolkit — AKI Prevention Toolkit. Intervention: All sites will receive the AKI Prevention Toolkit including 3 core interventions: 1. Standardized order sets; 2. IV and oral fluids; and 3. Reduced contrast volume. The interventions adhere to the KDIGO guidelines and add interventions developed and tested in our pilot intervention to implement AKI preventive strategies.
Behavioral: Technical Assistance (TA) — Technical Assistance (TA). Intervention: TA will be offered to the 8 teams randomized to the TA condition and will receive the AKI Prevention Toolkit plus monthly technical calls independently. TA arms will include TA with and without automated surveillance reporting (ASR).
  Arms: Technical Assistance (No ASR); Technical Assistance with ASR
Behavioral: Virtual Learning Collaborative (VLC) — Virtual Learning Collaborative (VLC). Intervention: The VLC will be offered to 8 teams and will receive the AKI Prevention Toolkit plus monthly virtual training calls with the other VLC sites. Each participating site will be supported to establish a multidisciplinary team charged with continuously improving AKI, which will include interventional cardiologists, cardiac catheterization lab manager and technicians, nursing representatives from the intensive care unit and/or holding areas, cardiology administration, nephrology, and representation from the quality improvement department (VA Clinical Application Coordinator [CAC] and Systems Redesign). VLC arms will include VLC with and without automated surveillance reporting (ASR).
  Arms: Virtual Learning Collaborative (No ASR); Virtual Learning Collaborative with ASR
Behavioral: Automated Surveillance Reporting (ASR) — Automated Surveillance Reporting (ASR). Intervention: The ASR will be offered to 8 teams. In addition to either TA or VLC, ASR teams will receive automated monthly reports in the form of an dashboard focused on AKI outcome and preventative measures overtime. The ASR report will be customized to each team and each individual operator and linked to their national VA-CART registry.
  Arms: Technical Assistance with ASR; Virtual Learning Collaborative with ASR

SUMMARY:
When a person has an imaging procedure that uses radio-contrast dye, there is a possibility of damage to that person's kidneys, which could result in being on dialysis or early death. The investigators are testing novel coaching and automated tools to help healthcare teams apply approaches that have been shown to prevent damage to kidneys during a cardiac catheterization procedure. The results of our study will help inform health care leaders on how to implement low-cost preventive strategies through team-based coaching and surveillance reporting for kidney injury and other patient safety priorities to every hospital in the United States.

DETAILED DESCRIPTION:
The investigators propose to test the implementation of evidence-based preventive interventions through a Virtual Learning Collaborative (VLC) with and without the novel use Automated Surveillance Reporting (ASR) intervention to change clinical practice and improve patient safety in common diagnostic procedures. Over 2 million people in the United States undergo diagnostic or interventional cardiac catheterization each year. Acute kidney injury (AKI), a patient safety metric set by the National Quality Forum, occurs in up to 14% of all patients following a procedure and up to 50% in patients with pre-existing chronic kidney disease (CKD), making AKI the most prevalent adverse event. Patients developing AKI have an increased risk of serious adverse events. There are widely accepted interventions to prevent AKI in patients undergoing cardiac catheterization. Our research team has demonstrated AKI can be prevented in 28% of patients with CKD through a large regional pilot. Our team has already developed ASR techniques for AKI nationally within the Veterans' Administration. Based on our own preliminary studies, the investigators hypothesize the incorporation of an automated plug-in ASR toolkit to provide near-realtime feedback to front-line care teams will significantly augment both VLC and Technical Assistance (TA) interventions in implementation trials. Our objective is to conduct a national randomized clinical trial testing the use of VLC or TA with or without a plug-in ASR toolkit to determine if ASR significantly improves outcomes for patients undergoing procedures with contrast dye to overcome the inconsistent application of known ways to prevent AKI. The rationale underlying the project is that ASR could prove to be a plug-in vehicle to improve patient endpoints in evidence-based preventive interventions in common diagnostic procedures. The investigators plan to test our hypothesis through the following specific aims in a 2x2 factorial cluster-randomized trial. For all aims, 16 hospitals will be randomized to receive one of the following interventions for 18-months: A) Technical Assistance (TA); B) Technical Assistance with Automated Surveillance Reporting (TA+ASR); C) Virtual Learning Collaborative (VLC) with team-based coaching (VLC); and D) Virtual Learning Collaborative with Automated Surveillance Reporting (VLC+ASR). Specific Aim 1: Compare the efficacy of a VLC and/or ASR compared to TA to reduce the incidence of AKI. Specific Aim 2: Evaluate the sustained efficacy of VLC and/or ASR to reduce the incidence of AKI following the intervention period. The interventions proposed use novel interactive video coaching sessions and ASR as low-cost scalable implementation strategies to prevent a clinical endpoint (AKI). Eighteen hospitals have agreed to participate and be randomized. The investigators expect the impact of a plug-in ASR to augment evidence based preventive interventions and VLC could significantly improve the consistent application of these interventions and implementation trials. In our opinion, our study will open the door to a new paradigm of implementation science seeking to continuously improve health care.

ELIGIBILITY:
Inclusion Criteria:

* VA Site Inclusion Criteria: All VA medical centers with a cardiac catheterization laboratory are eligible, and all catheterization operators at a site are included.
* Patient Inclusion Criteria: Among these sites, only patients aged 18 or greater with pre-existing CKD who undergo diagnostic coronary angiography or percutaneous coronary intervention (PCI or angioplasty) will be enrolled in the trial. CKD will be determined by a pre-existing CKD diagnosis in the VA medical record, or by two or more estimated glomerular filtration rates <60 (ml/min/1.73 m2) at least 90-days apart prior to presentation.

Exclusion Criteria:

* Patient Exclusion Criteria: Patients with a history of dialysis (hemodialysis, peritoneal dialysis), under the age of 18, or no evidence of pre-existing CKD will be excluded. Cardiac catheterization (also referred to as coronary angiography) is defined as a procedure in which a catheter is inserted into the femoral or radial artery and is threaded to the cardiac vasculature where radio-contrast dye is administered and a series of x-rays obtained in order to visualize the coronary arterial anatomy. PCI is when a clinical intervention is then performed to address any treatable pathology that is found.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10252 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremiah R Brown, PhD, Principal Investigator — Dartmouth College
Locations (2):
- United States (2):
  - Tennesee Valley VA, Nashville, Tennessee
  - White River Junction VA, White River Junction, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Tools (data, software, libraries, research tools, etc.) will be made available to all researchers in both the private and public sector free or for a nominal charge and with minimal restriction. An analytic program file used to produce the analyses and a de-identified dataset will be made available to third parties within the VA system to conduct confirmatory analyses for the proposed specific aims. All parties must be in compliance with VA regulations and access. All analytic program files (code) and results will be reported in supplementary appendixes for all publications.
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication and contingent on third party access to VA data and regulations.
Access Criteria: contingent on third party access to VA data and regulations

REFERENCES:
- [Derived] Matheny ME, Carpenter-Song E, Ricket IM, Solomon RJ, Stabler ME, Davis SE, Zubkoff L, Westerman DM, Dorn C, Cox KC, Minter FF, Jneid H, Currier JW, Athar SA, Girotra S, Leung C, Helton TJ, Agarwal A, Vidovich MI, Plomondon ME, Waldo SW, Aschbrenner KA, McKay V, O'Malley AJ, Brown JR. Sustained Improvements After Intervention to Prevent Contrast-Associated Acute Kidney Injury: A Randomized Controlled Trial. J Am Heart Assoc. 2025 May 20;14(10):e038920. doi: 10.1161/JAHA.124.038920. Epub 2025 May 15. PMID 40371586
- [Derived] Brown JR, Solomon R, Stabler ME, Davis S, Carpenter-Song E, Zubkoff L, Westerman DM, Dorn C, Cox KC, Minter F, Jneid H, Currier JW, Athar SA, Girotra S, Leung C, Helton TJ, Agarwal A, Vidovich MI, Plomondon ME, Waldo SW, Aschbrenner KA, O'Malley AJ, Matheny ME. Team-Based Coaching Intervention to Improve Contrast-Associated Acute Kidney Injury: A Cluster-Randomized Trial. Clin J Am Soc Nephrol. 2023 Mar 1;18(3):315-326. doi: 10.2215/CJN.0000000000000067. Epub 2023 Feb 8. PMID 36787125

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient procedures were excluded from analysis for one of three reasons: (1) missing post-operation creatinine, (2) history of prior dialysis, or (3) prior eGFR not meeting study eligibility criteria.
Units Other Than Participants: Hospitals
Groups:
- Virtual Learning Collaborative (No ASR): Virtual Learning Collaborative (VLC): The VLC will be offered to 10 teams and will receive the AKI Prevention Toolkit plus monthly virtual training calls with the other VLC sites. Each participating site will be supported to establish a multidisciplinary team charged with continuously improving AKI, which will include interventional cardiologists, cardiac catheterization lab manager and technicians, nursing representatives from the intensive care unit and/or holding areas, cardiology administration, nephrology, and representation from the quality improvement department (VA Clinical Application Coordinator [CAC] and Systems Redesign).
  AKI Prevention Toolkit: AKI Prevention Toolkit. Intervention: All sites will receive the AKI Prevention Toolkit including 3 core interventions: 1. Standardized order sets; 2. IV and oral fluids; and 3. Reduced contrast volume. The interventions adhere to the KDIGO guidelines and add interventions developed and tested in our pilot intervention to implement AKI preventive strategies.
- Virtual Learning Collaborative With ASR: Virtual Learning Collaborative (VLC): The VLC will be offered to 8 teams and will receive the AKI Prevention Toolkit plus monthly virtual training calls with the other VLC sites. Each participating site will be supported to establish a multidisciplinary team charged with continuously improving AKI, which will include interventional cardiologists, cardiac catheterization lab manager and technicians, nursing representatives from the intensive care unit and/or holding areas, cardiology administration, nephrology, and representation from the quality improvement department (VA Clinical Application Coordinator [CAC] and Systems Redesign). VLC arms will include VLC with and without automated surveillance reporting (ASR).
  AKI Prevention Toolkit: AKI Prevention Toolkit. Intervention: All sites will receive the AKI Prevention Toolkit including 3 core interventions: 1. Standardized order sets; 2. IV and oral fluids; and 3. Reduced contrast volume. The interventions adhere to the KDIGO guidelines and add interventions developed and tested in our pilot intervention to implement AKI preventive strategies.
  Automated Surveillance Reporting (ASR). Intervention: The ASR will be offered to 8 teams. In addition to either TA or VLC, ASR teams will receive automated monthly reports in the form of an dashboard focused on AKI outcome and preventative measures overtime. The ASR report will be customized to each team and each individual operator and linked to their national VA-CART registry.
Period: Overall Study
Arm/Group | Technical Assistance (No ASR) | Virtual Learning Collaborative (No ASR) | Technical Assistance With ASR | Virtual Learning Collaborative With ASR
Started | 2734; 5 Hospitals | 2967; 5 Hospitals | 2164; 4 Hospitals | 2387; 5 Hospitals
Completed | 830; 5 Hospitals | 1496; 5 Hospitals | 1073; 4 Hospitals | 1118; 5 Hospitals
Not Completed | 1904; 0 Hospitals | 1471; 0 Hospitals | 1091; 0 Hospitals | 1269; 0 Hospitals
Not completed — Ineligible for analysis | 1904 | 1471 | 1091 | 1269

BASELINE CHARACTERISTICS:
Population: Sites were randomized at the hospital level.
Units Other Than Participants: Hospitals
Groups:
- Total: Total of all reporting groups
Arm/Group | Technical Assistance (No ASR) | Virtual Learning Collaborative (No ASR) | Technical Assistance With ASR | Virtual Learning Collaborative With ASR | Total
Number analyzed (Participants) | 830 | 1496 | 1073 | 1118 | 4517
Number analyzed (Hospitals) | 5 | 5 | 4 | 5 | 19
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 70 [65 to 74] | 70 [63 to 74] | 70 [63 to 75] | 71 [64 to 75] | 70 [64 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 56 | 36 | 31 | 152
  Male | 801 | 1440 | 1037 | 1087 | 4365
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 110 | 371 | 316 | 161 | 958
  Race: Other | 46 | 72 | 71 | 124 | 313
  Race: White | 674 | 1053 | 686 | 833 | 3246

OUTCOME MEASURES:

1. Primary Outcome: Acute Kidney Injury
Description: Number of Participants with Acute Kidney Injury
Time Frame: within 48-hours of the procedure or within 7-days for in-patients, or onset of dialysis within 7-days
Measure: Count of Participants; unit: Participants
Arm/Group | Technical Assistance (No ASR) | Virtual Learning Collaborative (No ASR) | Technical Assistance With ASR | Virtual Learning Collaborative With ASR
Number analyzed (Participants) | 830 | 1496 | 1073 | 1118
Participants | 110 | 190 | 122 | 88

ADVERSE EVENTS:
Time Frame: 18-months
Arm/Group | Technical Assistance (No ASR) | Virtual Learning Collaborative (No ASR) | Technical Assistance With ASR | Virtual Learning Collaborative With ASR
All-Cause Mortality (participants affected / at risk) | 2/830 | 3/1496 | 1/1073 | 2/1118
Serious Adverse Events (participants affected / at risk) | 213/830 | 355/1496 | 331/1073 | 234/1118
Other Adverse Events (participants affected / at risk) | 0/830 | 0/1496 | 0/1073 | 0/1118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Technical Assistance (No ASR) (N=830) | Virtual Learning Collaborative (No ASR) (N=1496) | Technical Assistance With ASR (N=1073) | Virtual Learning Collaborative With ASR (N=1118)
New Onset Dialysis (Renal and urinary disorders) | 3 | 6 | 2 | 2
New Heart Failure (Cardiac disorders) | 79 | 162 | 127 | 91
Bleeding (Blood and lymphatic system disorders) | 17 | 24 | 50 | 20
Stroke (Vascular disorders) | 5 | 6 | 9 | 2
Myocardial Infarction (Cardiac disorders) | 109 | 157 | 143 | 119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT03556293/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT03556293/SAP_001.pdf